CLINICAL TRIAL: NCT04017195
Title: A Randomized, Double-blind, 2-Way Crossover Bioequivalence and Adhesion Study of a Transdermal Contraceptive Patch Manufactured With Newly Sourced Adhesive Components at the End of Shelf Life and Currently Marketed EVRA® at the Beginning of Shelf Life in Healthy Adult Women
Brief Title: A Study of New Transdermal Contraceptive Patch at End of Shelf Life and Currently Marketed EVRA at the Beginning of Shelf Life in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR108645; 2019-001893-27 (EudraCT Number); RWJ10553CON1019 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Sequence AB (Right/Left) (Experimental): A single patch of currently marketed EVRA patch using the adhesive component at the beginning of shelf life (BOSL) (Treatment A) will be applied to the right buttock of participants on Day 1 of Treatment Period 1, followed by application of a single patch of transdermal contraceptive using newly sourced adhesive component HMW PIB at the end of shelf life (EOSL) (Treatment B) to left buttock of participants on Day 1 of Treatment Period 2. The Treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: High molecular weight polyisobutylene (HMW PIB) patch (NGMN+EE) (Treatment B) (Test)
- Group 2: Sequence BA (Right/Left) (Experimental): Treatment B will be applied to the right buttock of participants on Day 1 in Period 1, followed by Treatment A to the left buttock on Day 1 in Period 2. The Treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: High molecular weight polyisobutylene (HMW PIB) patch (NGMN+EE) (Treatment B) (Test)
- Group 3: Sequence AB (Left/Right) (Experimental): Treatment A will be applied to the left buttock of participants on Day 1 in Period 1, followed by Treatment B to the right buttock on Day 1 in Period 2. The Treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: High molecular weight polyisobutylene (HMW PIB) patch (NGMN+EE) (Treatment B) (Test)
- Group 4: Sequence BA (Left/Right) (Experimental): Treatment B will be applied to the left buttock of participants on Day 1 in Period 1, followed by Treatment A to the right buttock on Day 1 in Period 2. The Treatment periods will be separated by a washout period of 21 days.
  Interventions: Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference); Drug: High molecular weight polyisobutylene (HMW PIB) patch (NGMN+EE) (Treatment B) (Test)

INTERVENTIONS:
Drug: EVRA patch (NGMN+EE) (Treatment A) (Reference) — A single transdermal contraceptive patch of EVRA (NGMN + EE) will be applied to the buttock (right or left) of participants on Day 1 of each Treatment period and is removed 7 days after patch application, that is, on Day 8.
  Other Names: RWJ10553
Drug: High molecular weight polyisobutylene (HMW PIB) patch (NGMN+EE) (Treatment B) (Test) — A single transdermal contraceptive HMW PIB (NGMN + EE) patch will be applied to the buttock (right or left) of participants on Day 1 of each Treatment period and is removed 7 days after patch application, that is, on Day 8.

SUMMARY:
The main objectives of this study are to determine the bioequivalence of the hormones (example, norelgestromin [NGMN] and ethinyl estradiol [EE]) from the transdermal contraceptive patch using the newly sourced adhesive component as compared to the currently marketed EVRA patch using the adhesive component, evaluate the adhesion of the transdermal contraceptive patch using the newly sourced adhesive component as compared to the currently marketed EVRA patch using the adhesive component and show non-inferior adhesion of the transdermal contraceptive patch using the newly sourced adhesive component as compared to the currently marketed EVRA patch using the adhesive component.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2), inclusive, and body weight not less than 50 kilogram (kg) and not more than 100 kg at screening
* Participant must be surgically sterile with intact ovaries, abstinent, or, if sexually active, be practicing a highly effective method (that is, failure rate of less than [<] 1 percent [%] per year) of non hormonal contraception (example, intrauterine device [IUD], male partner sterilization) before admission and throughout the study
* Participant has a blood pressure (after the participant is supine or sitting for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Participant must have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: Normal sinus rhythm with heart rate between 45 and 100 beats per minute (bpm), extremes included; QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) =<470 millisecond (ms); QRS interval =<120 ms; PR interval =<220 ms. ECG morphology consistent with healthy cardiac conduction and function. Any evidence of heart block and left or right bundle branch block is exclusionary
* Participant must be a non-smoker, ex-smoker for greater than (>) 6 months, must not use nicotine containing substances including tobacco products (example, cigarettes, e-cigarettes. cigars, chewing tobacco, gum, patch), or tests negative for cotinine at screening and on Day 1 of each treatment period

Exclusion Criteria:

* Participant has clinically significant abnormal values for hematology, biochemistry, or urinalysis at screening as deemed appropriate by the investigator
* Participant has abnormal thyroid stimulating hormone level at screening
* Participant has evidence of cervical dysplasia as documented by a CytoRich test or Papanicolaou (PAP) smear test within 10 months before screening. If a PAP smear has been done within 10 months prior to screening and results are available (documentation is available at the study site) a cervical smear does not need to be performed
* Participant has used oral hormonal contraception, that is, contraceptive pills, within 3 months before admission to the study site on Day -1 of Treatment Period 1
* Participant currently has a contraceptive implant such as Implanon or Norplant in place, or has had removal of contraceptive implant within the 3 months before admission to the study site on Day -1 of Treatment Period 1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Mean Steady-State Concentration (Css) of Norelgestromin (NGMN) | 48 to 168 hours post-dose
  Css is the mean steady-state concentration for NGMN after patch application, will be calculated, as the mean concentration between 48 hours and 168 hours, inclusive, after patch application.
Mean Steady-State Concentration (Css) of Ethinyl Estradiol (EE) | 48 to 168 hours post-dose
  Css is the mean steady-state concentration for EE after patch application, will be calculated, as the mean concentration between 48 hours and 168 hours, inclusive, after patch application.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of NGMN | Predose, 24, 48, 72, 96, 120, 144, 168, 168.5, 171, 174, 180, 192, 216 and 240 hours post dose
  Tmax is the time to reach the maximum observed plasma concentration of NGMN will be assessed.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of EE | Predose, 24, 48, 72, 96, 120, 144, 168, 168.5, 171, 174, 180, 192, 216 and 240 hours post dose
  Tmax is the time to reach the maximum observed plasma concentration of EE will be assessed.
Area Under the Plasma Concentration-Time Curve from Time 0 (Patch Application) to Time 168 hours Post-dose (AUC[0-168]) of NGMN | Pre-dose to 168 hours post-dose
  AUC(0-168) is the area under the concentration versus time curve from zero (patch application) to 168 hours of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 168 hours Post-dose (AUC[0-168]) of EE | Pre-dose to 168 hours post-dose
  AUC(0-168) is the area under the concentration versus time curve from zero (patch application) to 168 hours of EE in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 240 hours Post-dose (AUC[0-240]) of NGMN | Pre-dose to 240 hours post-dose
  AUC(0-240) is the area under the concentration versus time curve from zero (patch application) to 240 hours of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Time 240 hours Post-dose (AUC[0-240]) of EE | Pre-dose to 240 hours post-dose
  AUC(0-240) is defined as area under the concentration versus time curve from zero (patch application) to 240 hours of EE in plasma will be assessed.
Cumulative Adhesion Percentage Ratio | Baseline (Day 1) and every 24 hours after patch application up to patch removal at 168 hours (Day 8)]
  Adhesion of patches will be assessed in accordance with the European Medicines Agency (EMA) 0-5 scoring system. An estimated percentage of adhesion, to a whole integer, will be obtained (EMA 0-5 [percentage (%)] scoring). Estimated percentages of adhesion and corresponding EMA 0-5 score at each interval will be recorded in each participant's electronic case report form. The scoring system for adhesion of transdermal patches is indicated as follows : 0= greater than (>) 90-100% of the patch area adheres; 1= >80-90% of the patch area adheres; 2= >70-80% of the patch area adheres; 3= >60-70% of the patch area adheres; 4= >50-60% of the patch area adheres; 5= 0-less than or equal to (<=) 50% of the patch area adheres.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Infinite Time (AUC[0-infinity]) for NGMN | Pre-dose to 240 hours post-dose
  AUC (0-infinity) is the area under the concentration versus time curve from zero (patch application) to infinite time of NGMN in plasma will be assessed.
Area Under the Plasma Concentration-Time Curve From Time 0 (Patch Application) to Infinite Time (AUC[0-infinity]) for EE | Pre-dose to 240 hours post-dose
  AUC (0-infinity) is the area under the concentration versus time curve from zero (patch application) to infinite time of EE in plasma will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants with Specific Application Site Reactions | Pre-dose, 168.5, and 192 hours post-dose
  Percentage of participants with specific application site reactions (including erythema, edema, pustules, papules and itching) will be summarized for each treatment.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 97 Days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- SGS Belgium NV, Antwerp, Belgium
- Charite - Universitaetsmedizin Berlin (CCM), Berlin, Germany
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency